CLINICAL TRIAL: NCT00493779
Title: An Exploratory, Multi-Center, Open-Label, Single-Arm Study to Evaluate the Discontinuation Effect of Clopidogrel After Drug Eluting Stent (DECADES) on Inflammatory and Platelet Activation Markers in Subjects Who Are Receiving Low Dose Acetylsalicylic Acid (ASA)
Brief Title: A Study to Evaluate the Discontinuation Effect of Clopidogrel After Drug Eluting Stent Implantation in Non-diabetic Patients
Acronym: DECADES
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: CV149-208; Eudract number: 2007-000713-11
Record Dates: First submitted 2007-06-27; First posted 2007-06-28 (Estimated); Results first posted 2009-08-11 (Estimated); Last update posted 2010-08-10 (Estimated); Status verified 2010-06

CONDITIONS: Antiplatelet Aggregation
MeSH Terms: interventions — Blood Specimen Collection

ARMS (1):
- 1 (No Intervention): Effect of Clopidogrel withdrawal on biomarkers will be assessed via blood draws
  Interventions: Procedure: Blood Collection

INTERVENTIONS:
Procedure: Blood Collection — 4 weeks

SUMMARY:
The purpose of the study is to look at the biomarkers of inflammation and platelet activation in patients with drug eluting stents implanted approximately 12 months ago on aspirin and statin, for a 4-week period after the routine discontinuation of clopidogrel

ELIGIBILITY:
Inclusion Criteria:

* Subjects with one or more drug-eluting stents of any type who are coming to the end of their 12 months of clopidogrel (75 mg daily) treatment
* Subjects receiving low dose ASA
* Subjects receiving a statin
* Current medication regimen (including ASA and statins) must have been stable for three (3) months. i.e. no initiation of new prescription medication or change in dosage of any previously initiated medication within three (3) months of entering this study
* Subjects with no clinical history of diabetes mellitis
* Men and women, ages 18 years or older

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2007-10; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (6):
- Local Institution, Paris, France
- Local Institution, Mainz, Germany
- Netherlands (2):
  - Local Institution, Nieuwegein
  - Local Institution, Rotterdam
- United Kingdom (2):
  - Local Institution, Glasgow, Central
  - Local Institution, Southampton, Hampshire

REFERENCES:
- [Background] Wykrzykowska JJ, Warnholtz A, de Jaeger P, Curzen N, Oldroyd KG, Collet JP, Ten Berg JM, Rademaker T, Goedhart D, Lissens J, Kint PP, Serruys PW. Effect of clopidogrel discontinuation at 1 year after drug eluting stent placement on soluble CD40L, P-selectin and C-reactive protein levels: DECADES (Discontinuation Effect of Clopidogrel After Drug Eluting Stent): a multicenter, open-label study. J Thromb Thrombolysis. 2009 Nov;28(4):410-7. doi: 10.1007/s11239-009-0354-y. PMID 19504052

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 103 subjects who were enrolled and treated with clopidogrel, were enrolled, of which 98 subjects had discontinued clopidogrel treatment and entered follow-up phase (study phase).
Groups:
- Clopidogrel Withdrawal Population: All enrolled participants in whom clopidogrel treatment was discontinued.
Period: Overall Study
Arm/Group | Clopidogrel Withdrawal Population
Started | 98 (Number of subjects who had discontinued clopidogrel treatment and entered follow-up phase)
Completed | 97 (Completed follow-up phase)
Not Completed | 1
Not completed — Logistical issue at site | 1

BASELINE CHARACTERISTICS:
Arm/Group | Clopidogrel Withdrawal Population
Number analyzed (Participants) | 98
Age Continuous [Mean (Standard Deviation); unit: years] | 63.3 (8.5)
Age Continuous [Median (Full Range); unit: years] | 63 [44 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 78
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 93
  Asian Oriental | 5
Mean Baseline High Sensitivity C-Reactive Protein (hs-CRP) [Mean (Standard Deviation); unit: mg/L] | 1.70 (2.052)
Mean Baseline Plasma Soluble P-Selectin [Mean (Standard Deviation); unit: ng/mL] | 44.59 (14.898)
Mean Baseline Soluble CD40 Ligand [Mean (Standard Deviation); unit: ng/L] | 223.76 (186.513)

OUTCOME MEASURES:

1. Secondary Outcome: Adjusted Mean Percent Changes From Baseline in Plasma Soluble P-Selectin
Description: Based on ANCOVA models performed on log scale controlling for site and natural logarithm of baseline Plasma Soluble P-selectin value. Percent changes from baseline can be interpreted as difference of biomarker timepoint value minus baseline value divided by baseline value. Positive percent change is known to be mediated by increases in sCD40L.
Time Frame: Week 1, Week 2, Week 3, Week 4
Population: Number of patients in the biomarker analysis population having baseline Plasma Soluble P-selectin value (n=95) and at least one post-clopidogrel withdrawal measurement for Plasma Soluble P-selectin value. No imputation technique for missing values was applied.
Measure: Mean (Standard Error); unit: percent change
Groups:
- Biomarker Analysis Population: All participants in the Clopidogrel Withdrawal Population having a baseline and at least one post clopidogrel withdrawal measurement for any of the 3 biomarkers collected.
Arm/Group | Biomarker Analysis Population
Number analyzed (Participants) | 95
percent change
  Baseline Value (units=ng/mL) (n=95) | 44.59 (1.53)
  Mean Percent Change from Baseline at Week 1 (n=92) | 9.00 (2.38)
  Mean Percent Change from Baseline at Week 2 (n=91) | 11.10 (2.11)
  Mean Percent Change from Baseline at Week 3 (n=91) | 3.63 (2.69)
  Mean Percent Change from Baseline at Week 4 (n=89) | 1.90 (2.76)

2. Primary Outcome: Adjusted Mean Percent Changes From Baseline in Soluble CD40 Ligand (sCD40L)
Description: Based on ANCOVA models performed on log scale controlling for site & natural logarithm of baseline soluble CD40 Ligand value. Percent changes from baseline can be interpreted as the difference of biomarker timepoint value minus baseline value divided by baseline value. Positive percent change might indicate possible enhanced platelet activation.
Time Frame: Week 1, Week 2, Week 3, Week 4 (primary timepoint)
Population: Number of participants in the biomarker analysis population having a baseline soluble CD40 Ligand value (n=95) and at least one post-clopidogrel withdrawal measurement for soluble CD40 Ligand value. No imputation technique for missing values was applied.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Biomarker Analysis Population
Number analyzed (Participants) | 95
percent change
  Baseline value (units=ng/L) (n=95) | 223.76 (19.14)
  Mean Percent Change from Baseline at Week 1 (n=92) | 35.04 (10.37)
  Mean Percent Change from Baseline at Week 2 (n=91) | 38.88 (10.76)
  Mean Percent Change from Baseline at Week 3 (n=91) | 32.74 (9.68)
  Mean Percent Change from Baseline at Week 4 (n=89) | 39.42 (11.07)

3. Secondary Outcome: Adjusted Mean Percent Changes From Baseline in Hs-CRP
Description: ANCOVA models performed on log scale controlling for site & natural logarithm of baseline hs-CRP. Back-transformed mean percent changes are presented. Percent changes from baseline can be interpreted as difference of biomarker timepoint value - baseline value ÷ baseline value. Since there is no measure of platelet inhibition or overall thrombogenicity assay presented here, a negative percent change for this measure can not be judged on its own as indicating improvement.
Time Frame: Week 1, Week 2, Week 3, Week 4
Population: Number of patients in the biomarker analysis population having baseline hs-CRP value and at least one post clopidogrel withdrawal measurement for hs-CRP value. No imputation technique for missing values was applied.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Biomarker Analysis Population
Number analyzed (Participants) | 98
percent change
  Baseline Value (units=mg/L) (n=98) | 1.70 (0.21)
  Mean Percent Change from Baseline at Week 1 (n=97) | -20.59 (6.76)
  Mean Percent Change from Baseline at Week 2 (n=95) | -22.89 (6.78)
  Mean Percent Change from Baseline at Week 3 (n=96) | -19.32 (8.22)
  Mean Percent Change from Baseline at Week 4 (n=96) | -17.70 (8.48)

4. Secondary Outcome: Adverse Events (AE) / Serious Adverse Events (SAE)Deaths, and AEs Leading to Discontinuation of Follow-up
Description: An AE is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a patient or clinical investigation subject administered an investigational (medicinal) product and that does not necessarily have a causal relationship with this treatment. An SAE is any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is an important medical event.
Time Frame: Throughout 4-week follow-up period
Population: All enrolled patients in whom clopidogrel treatment was discontinued.
Measure: Number; unit: Participants
Arm/Group | Clopidogrel Withdrawal Population
Number analyzed (Participants) | 98
Participants
  Deaths | 0
  Any AE | 20
  AEs leading up to Discontinuation | 0
  SAEs | 2

ADVERSE EVENTS:
Arm/Group | Clopidogrel Withdrawal Population
Serious Adverse Events (participants affected / at risk) | 2/98
Other Adverse Events (participants affected / at risk) | 0/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Clopidogrel Withdrawal Population (N=98)
Non-cardiac chest pain (General disorders) | 1
Angina unstable (Cardiac disorders) | 1

LIMITATIONS AND CAVEATS:
The open-label and exploratory nature of this small study and the absence of control group inherently limit the interpretability of the results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.